CLINICAL TRIAL: NCT06335108
Title: Prospective Unicentre Non-randomised Study: Comparison of Postoperative Pain After Breast Cancer-typical Surgery Under Tumescent Local Anaesthesia Versus General Anaesthesia - TLA 001
Brief Title: Postoperative Pain After Breast Surgery Under Tumescent Local Anaesthesia Versus General Anaesthesia ( TLA-001 )
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: SenoEx_TLA_Maligne
Record Dates: First submitted 2024-03-12; First posted 2024-03-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma; Breast Carcinoma in Situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Surgery carried out according to clinical routine under general anaesthesia.
  Interventions: Procedure: General Anaesthesia
- Local Anaesthesia Group: Surgery carried out under local tumescent anaesthesia. Procedure
  Interventions: Procedure: Local tumescent anaesthesia

INTERVENTIONS:
Procedure: General Anaesthesia — Breast surgery is carried out under general anesthesia.
  Groups: Control Group
Procedure: Local tumescent anaesthesia — Breast surgery is carried out under local tumescent anesthesia.
  Groups: Local Anaesthesia Group

SUMMARY:
The present study aims to investigate the impact of Tumescent Local Anesthesia (TLA) on pain perception following surgeries typical for breast cancer. Previous research has already confirmed the feasibility of conducting operations in TLA for benign breast conditions. In contrast to general anesthesia, Tumescent Local Anesthesia involves local anesthesia of the surgical site, allowing patients to remain awake during the procedure and eliminating the risks associated with general anesthesia. Additionally, if needed, sedatives or further anesthesia can be administered through the vein. Building upon the successful applications of TLA in benign breast surgeries, this follow-up study at the Department of Women's Health focuses on enhancing surgical techniques, pain management, and postoperative care for breast cancer-related procedures. Simultaneously, our goal is to gather scientific data regarding the application of this technique. This research contributes to the continuous advancement of medical practices in the field of breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Written informed consent
* Histologically confirmed breast carcinoma or pure ductal carcinoma in situ
* Planned operation:
* Segmental resection/ breast-conserving surgery
* Segmental resection/ breast-conserving surgery with SNB
* Ablatio
* Ablatio with SNB/ axilla exploration

Exclusion Criteria:

* Expected lack of patient compliance or inability of the patient to understand the purpose of the study
* Lack of patient consent
* Pregnancy
* Complete axillary dissection
* Tumour-adapted reduction surgery, implant reconstructions
* Surgeries where technical difficulties are expected under any anaesthesia (e.g. ASA IV, BMI > 40)
* Bilateral breast operations
* Men

Exclusion Criteria for surgery in TLA:

* Injection phobia
* Psychoses/ previous psychological illnesses
* Advanced dementia
* Language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients presenting with invasive breast carcinoma or pure ductal carcinoma in situ with an indication for surgical treatment at the Department of Women's Health in Tübingen.
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 5 weeks
  The primary endpoint is the recording of postoperative pain. Pain will be measured on 1.-3. postoperative day using the Visual Analogue Scale (VAS). The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
  Additionally, the postoperative pain will be assessed using the VAS at the post-operative follow-up consultation, which usually takes place 2-5 weeks after surgery.

SECONDARY OUTCOMES:
HRQoL/ Quality of life | 5 weeks
  The outcome measure for Health-Related Quality of Life (HRQoL) in this study utilizes the Breast-Q questionnaire specific to breast cancer (BCT/Mastectomy). Preoperative assessments are conducted during the recruitment phase following participants' consent, providing baseline HRQoL data. Postoperative evaluations occur 2-5 weeks after the surgery during follow-up discussions, capturing changes in HRQoL in the immediate aftermath of the mastectomy and informing the study about the impact of the surgical intervention on participants' quality of life.
Postoperative pain medication requirements | 5 weeks
  The outcome measure for postoperative pain medication requirements includes the assessment of administered pain medications, encompassing anti-inflammatory drugs, opioids, and non-opioid analgesics.
  Patient's medical records will be examined to identify the pain medications administered postoperatively. The administered pain medications will then be categorized into anti-inflammatory drugs, opioids, and non-opioid analgesics. The total dosage of each type of pain medication administered will be calculated until hospital dischanrge. To evaluate the effectiveness of the administered pain medications in managing postoperative pain, pain assessment tool (Visual Analog Scale) will be used to measure pain intensity (2-3x daily for exercise and rest). On the first postoperative day, patients also receive the standardized QUIPS pain questionnaire consisting of 16 questions pain assesement after operation.
Complications | 5 weeks
  Complications in the study will be recorded during the hospital stay and post-operative follow-up, using the Clavien- Dindo classification system to categorize and assess their severity, contributing vital insights into the safety and efficacy of the surgical intervention.
Length of hospital stay | 1 day until 2 weeks
  The "length of hospital stay" refers to the time elapsed from a patient's admission to their discharge.
Duration of surgery | 1 until 5 hours
  In the current clinical study, the duration of surgery, measured as the time from incision to wound closure, will be meticulously recorded using precise timekeeping instruments. This involves capturing the elapsed time from the moment the surgical incision is made to the point when the wound is closed.
Drainage delivery rate | Surgery until discharge (1 day until 2 weeks )
  The drainage delivery rate will be assessed by measuring the volume of fluid collected by the drainage system until the point of discharge. This involves tracking the total volume in milliliters (ml) accumulated over the entire duration of drainage until the patient is discharged.
Follow-up surgery for R1 situation | 5 hours
  An additional outcome criterion is whether there is a R1 situation with subsequent surgery, answered yes/no.
Preoperative fear of surgery and anaesthesia | 30 Minutes
  The secondary outcome criterion, "preoperative fear of surgery and anesthesia," will be assessed using the APAIS (Amsterdam Preoperative Anxiety and Information Scale) questionnaire and a Visual Analog Scale (VAS) ranging from 0 to 10. The APAIS questionnaire consists of multiple items measuring anxiety and information desire related to surgery and anesthesia, with higher scores indicating greater preoperative fear. The Visual Analog Scale, ranging from 0 (no fear) to 10 (extreme fear), allows participants to subjectively rate their apprehension, providing a numerical representation of the intensity of preoperative fear.
Costs | 5 weeks
  The costs of breast surgery conducted under general anesthesia versus local anesthesia serve as a crucial outcome criterion in the clinical study. This assessment involves comparing the overall expenses associated with each anesthesia method, including anesthesia administration, recovery, and potential complications, to determine the economic implications and cost-effectiveness of the two approaches in the context of breast surgery.
Satisfaction of the surgeon with the course of the operation | 5 hours
  The satisfaction of the surgeon with the course of the operation will be measured on a scale of 0 to 10, where 0 represents not satisfied at all and 10 signifies extreme satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Böer, Dr., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Women's Hospital, Tübingen, Germany